CLINICAL TRIAL: NCT04859374
Title: Effectiveness of Home- Behavioral Approach by Mindfulness Added to Pharmacological Treatment on Endogenous Pain Modulation in Patients With Chronic Pain: Results at Long-term (Be-Home-Pain)
Brief Title: Chronic Pain and Conditioned Pain Modulation After on Line-behavioral Approach
Acronym: Be-Home-Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Be-Home-Pain
Record Dates: First submitted 2021-03-31; First posted 2021-04-26 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-04

CONDITIONS: Migraine
Keywords: Chronic Pain;; Chronic Migraine;; Conditioned Pain Modulation;; Mindfulness;
MeSH Terms: conditions — Migraine Disorders; Chronic Pain | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (TAU) (Other): Any pharmacological therapy used for managing chronic pain or chronic migraine
  Interventions: Drug: treatment as usual (TAU) (pharmacological)
- TAU plus behavioral approach (Other): Any pharmacological therapy used for managing chronic pain or chronic migraine added with behavioral approach (mindfulness) delivered on line and smart phone for 6 weekly sessions
  Interventions: Behavioral: Mindfullness; Drug: treatment as usual (TAU) (pharmacological)

INTERVENTIONS:
Behavioral: Mindfullness — Behavioral approach (mindfulness) delivered on line and smart phone for 6 weekly sessions
  Arms: TAU plus behavioral approach
Drug: treatment as usual (TAU) (pharmacological) — Any pharmacological therapy used for managing chronic pain or chronic migraine

SUMMARY:
Chronic pain is a disabling condition associated with progressive changes and decline in psychological wellbeing. According with a modern conceptualization, pain has to be considered a biopsychosocial disorder where biological, affective, social and psychological aspects are strictly connected. Although this new conceptualization, the implementation of an integral systems approach of psychological tenets into treatments for chronic pain are limited. Concerning treatments of chronic pain condition, the literature of the last years has demonstrated how clinical benefit can be improved when traditional therapies are combined with behavioral approaches in particular mindfulness. Systemic quantitative-somatosensory testing of Conditioned Pain Modulation (CPM) can be considered a measure of endogenous modulation of pain and it has been used in different clinical experiences to evaluate the effectiveness of different pain treatments even if non pharmacological approaches.

DETAILED DESCRIPTION:
Chronic pain is a disabling condition associated with progressive changes and decline in psychological wellbeing. The burden of this condition is significant and also the epidemiological impact. According with a modern conceptualization, pain has to be considered a biopsychosocial disorder where biological, affective, social and psychological aspects are strictly connected. Although this new conceptualization, the implementation of an integral systems approach of psychological tenets into treatments for chronic pain are limited. Concerning treatment of chronic pain condition, the literature of the last years has demonstrated how clinical benefit can be improved when traditional therapies are combined with behavioral approaches in particular mindfulness, that help patients to become more conscious about their symptoms and able to manage pain without medication.

Systemic quantitative-somatosensory testing of Conditioned Pain Modulation (CPM) can be considered a measure of endogenous modulation of pain and it has been used in different clinical experiences to evaluate the effectiveness of different pain treatments even if non pharmacological approaches Aim of this study: A group of patients suffering from Chronic Migraine and Chronic Neuropathic Pain will be studied and followed with a specific mindfulness protocol, added to traditional pharmacological therapy, performed on-line for 8 weeks. In order to determine if the behavioral approach can improve their clinical condition patients will be followed for 12 months after treatments with regular visits every 3 months.

Also, in order to assess the integrity and improvement of the endogenous pain inhibitory control a conditioned pain modulation paradigm will be performed at baseline and at 3, 6, 12 months. Patients will perform a baseline evaluation of thermal pain and mechanical pain tresholds using the quantitative sensory methods, including the determination of heat-generated temporal summation. Then, at baseline and at 3, 6, 12 months follow up, the CPM paradigm will be performed using two heat painful stimuli, a tonic heat stimulus as conditioning stimulus and a phasic heat stimulus as test stimuli.

Patients will be treated by traditional pharmacological therapies added to behavioral approach (mindfulness on line by using a specific platform (STARLEAF)) (TAU/MIND) Eight weekly one-hour video-sessions of mindfulness practice will be scheduled for patients; instructions to manage pain and to encourage the use of strategies for pain management will be given.

Moreover, instructions for behavioral approach and mindfulness, to practice every day will be given: daily standardized mindfulness sessions of 12 minutes, by smartphone, recorded by the expert who generally manages their sessions at the hospital will be scheduled for patients Neuropsychological assessment will be provided at baseline and at every follow up Clinical, neurophysiological and neuropsychological results will be compared to those obtained from another group of patients treated by traditional pharmacological treatment (TAU) This preliminary study will be conducted on 35 patients with diagnosis of CM and Chronic Neuropathic Pain performed at our center.

Specific questionnaires for cognitive assessment and disability, catastrophizing attitude, anxiety, depression, acceptance, pain coping will be performed at baseline and repeated at every follow up ( PCS; GSE; HADS; CPAQ; AAQ; MAAS). The pain diary will be checked too with scheduled NSR evaluation. The questionnaires will be repeated at every follow up and the pain diary will be evaluated.

Results will be collected at baseline up to 12 months after treatment for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic Migraine and Chronic Neuropathic Pain
* Written informed consent

Exclusion Criteria:

* Co-existent severe medical or psychiatric illnesses
* Use of opioids during the 3 months before the inclusion into the protocol
* Practice of mindfulness in the last 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Change of pain intensity | From the first visit to the first follow up at 3 months till the last follow up at 12 months
  Mean NRS (Numerical Rating Scale evaluation from the Daily diary card ) difference of at least 2 points on the scale(the scale range is from 0=no pain to 10 =maximum pain perceived) between MIND/TAU and TAU groups assessed by the daily diary card.

SECONDARY OUTCOMES:
Change of pain frequency | 6 and 12 months
  Decrease in pain frequency, (days of pain per month) assessed by Daily Diary Card.
Change of medication intake | 6 and 12 months
  Decrease of number of symptomatic medications per month assessed by Daily Diary Card.
Neurophysiological indexes | 3, 6 and 12 months
  Changes in neurophysiological indexes evaluated by quantitative sensory test for conditioned pain modulation analysis.
Psychological measures - coping strategies | 6 and 12 months
  * Pain Catastrophizing Scale-Italian, PCS-I (Monticone et al., 2012)
  * cut-off: 0 - 30 normal ranges > 30 abnormal
Psychological measures - Quality of life | 6 and 12 months
  * General Self-Efficacy Scale, GSE ( (Schwarzer et al., 1995)
  * cut off: 0 - 10 abnormal 10 - 40 normal ranges
Psychological measures - Mood | 6 and 12 months
  * Hospital Anxiety and Depression Scale, HADS (Costantini et al., 1999)
  * cut-off: total score 0 -7 = normal total score > 7 = impairment
Psychological measures - Mindfulness specific tests | 6 and 12 months
  * Mindful Awareness Attention Scale, MAAS (Veneziani et al., 2015) for mindfulness attitude for patients randomized in the MIND/TAU group
  * cut-off: 15 - 90 normal ranges

IPD SHARING:
Plan to Share IPD: No